CLINICAL TRIAL: NCT03822299
Title: Effects of Faecal Microbiota Transplantation in Patients With Irritable Bowel Syndrome: A Randomised, Double-blind Placebo-controlled Study
Brief Title: Effects of Faecal Microbiota Transplantation in Patients With IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Fonna (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Principal Investigator, Magdy El-Salhy, MD, PhD, Professor/Consultant gatroenterologist, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HelseFonna
Record Dates: First submitted 2018-12-21; First posted 2019-01-30 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention. Dietary supplement: fecal suspension. Healthy donor or own faeces (placebo) administrated through working canal of a gastroscope.
Who Masked: Outcomes Assessor
Masking Description: A research nurse, not involved in the trial, create the allocation sequence using a website. This was done in blocks of 21 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (No Intervention): Patients receive suspension of their own feces.
- 30 g donor dose (Active Comparator): Patients receiving 30 g of a healthy donor feces.
  Interventions: Dietary Supplement: healthy feces microbiota
- 60 g donor dose (Active Comparator): Patients receiving 60 g of a healthy donor feces.
  Interventions: Dietary Supplement: healthy feces microbiota

INTERVENTIONS:
Dietary Supplement: healthy feces microbiota — Suspension of healthy feces microbiota in sterile saline solution
  Other Names: placebo
  Arms: 30 g donor dose; 60 g donor dose

SUMMARY:
Irritable bowel syndrom (IBS) is a common chronic gastrointestinal disorder that affects 10-20% of the world population. The prevalence of IBS in Norway is between 8% and 25%. The pathophysiology of IBS is incompletely understood, and there is no effective treatment for this condition. Imbalance (dysbiosis) of the gut microbiome has been found in patients with IBS. In the absence of effective method to restore the dysbiosis, transplantation of a microbiome from healthy individuals with well-functioning gut (FMT) to those with IBS has been performed. Two randomized double blind placebo-controlled (RCT) studies have been published recently. Whereas it was reported in one study that FMT reduced symptom and improved quality of life in patients with IBS, FMT had no effect in the other study. In order to clarify these contradictory results, a new RCT study that enrolled larger number of patients is required. In this study, the investigators intend to recruit 170 IBS patients from those attending outdoor clinic at Stord hospital in a randomized, double blind placebo trial. A single healthy donor with well-characterized microbiome is going to be used. The effects on symptoms, quality of life, fatigue as well as dysbiosis before and after FMT are going to be investigated. The possible mechanisms behind the effects if any of FMT such as changes in intestinal stem cells, enteroendocrine cells and local immune defense shall be also investigated. The patients are going to be randomized either to placebo (own faces), 30 g or 60 g of the donor faces in ratio 1:1:1.

DETAILED DESCRIPTION:
Study design Patients One hundred and seventy patients who fulfill the following inclusion criteria and lack the exclusion criteria shall be included. In addition, the patients are examined physically, and blood tests are taken to exclude inflammation, and liver, kidney and thyroid diseases. They undergo further gastroscopy with duodenal biopsies to exclude coeliac disease. They undergo also colonoscopy to exclude malignity, or inflammatory bowel disease (IBD). Microscopic colitis is excluded by examining tissue obtained by colonoscopy with segmental biopsy sampling.

Donor selection and screening:

A single donor shall be selected and screened according to the European and international guidelines. The donor should not be a first-degree relative to any of the patients, as the intestinal microbiota is affected by the genetic composition, and similarity between the donor and recipient in the fecal microbiota may occur.

Protocol

Feces collection, preparation and administration:

Feces from both the donors and recipients were collected and stored at - 80•. Frozen feces (30 or 60g) from the donor or patients (placebo), thawed at 5° C and were dissolved in 50 mL of 0.9% sterile saline per 30 g feces. The dissolved stool is administrated to the patients, after overnight fast, through working channel of gastroduodeno-scope in pars descendent duodenum distal to the papilla of Vater.

Sigmoidoscopy: After administration of faeces, a sigmoidoscopy is performed during which 4 biopsies from the sigmoid colon about 30 cm from anus, and 4 biopsies from the rectum about 15 cm from anus are taken. Sigmoidoscopy is repeated in the same way 1 month after FMT.

Methods Questionnaires

1. IBS symptom severity Scale (IBS-SSS) questionnaire.
2. Birmingham Symptom scale questionnaires.
3. IBSQoL questionnaire.
4. Short form of Nepean Dyspepsia Index (SF-NDI) questionnaire.
5. Fatigue Assessment Scale (FAS).

Microbiome analysis Gut microbiota analysis was performed using the GA-mapTM Dysbiosis test (Genetic Analysis AS, Oslo, Norway) by algorithmically assessing fecal bacterial abundance and profile (dysbiosis index, DI), and potential deviation in the microbiome from normobiosis. GA-map test is based on fecal homogenization, mechanical bacterial cell disruption and automated total bacterial genomic DNA extraction using magnetic beads. DI is based on 54 DNA probes targeting more than 300 bacterial strains based on their 16S rRNA sequence in seven variable regions (V3-V9). Twenty-six bacteria probes are species specific, 19 detect bacteria on genus level, and 9 probes detect bacteria at higher taxonomic levels. Probe labeling is by single nucleotide extension and hybridization to complementary probes coupled to magnetic beads, and signal detection by using Bio Code 1000A 128-Plex Analyzer (Applied Bio Code, Santa Fe Springs, CA, USA). A DI above 2 shows a microbiota profile that differs from that of the normobiotic reference collection (DI 1-2: non-dysbiosis, DI: moderate, DI 4-5: severe dysbiosis).

ELIGIBILITY:
Inclusion criteria:

1. Patients between who fulfill Rome IV criteria for the diagnosis of IBS.
2. Patients with moderate to severe IBS symptoms (IBS-SSS ≥ 175).

Exclusion criteria:

1. Pregnant, planning pregnancy or lactating women.
2. The use of antibiotics or probiotics within 1 month prior to FMT.
3. Patients who had undergone any abdominal surgery, with the exception of appendectomy, cholecystectomy, Caesarean section or hysterectomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Global improvement in IBS symptoms as assessed by IBS Symptom Severity Scale (IBS-SSS) | 3 months.
  IBS-SSS is a visual assessment scale (VAS) rating from 0 to 100, with total scores ranging from 0 to 500. Lower scores indicate improvement.
Global improvement in IBS symptoms as assessed by Birmingham Symptom scale questionnaire | 3 months.
  This questionnaire consists of 11 question. measured on a six-point Likert scale ranging from 0 to 5. Lower scores indicate improvement.
Quality of life as assessed by IBS quality of life (IBSQoL) questionnaire | 3 months
  IBSQoL consist of 34- questions measured on a five-point Likert scale ranging from 0 to 5. Higher scores indicate improvement.
Quality of life as assessed by Short form of Nepean Dyspepsia Index (SF-NDI) questionnaires | 3 months
  SF-NDI is a five-point Likert scale ranging from 0 to 5. Lower scores indicate improvement.
Fatigue as assessed by: Fatigue Assessment Scale (FAS) questionnaire | 3 months
  FAS is a five-point Likert scale ranging from 0 to 5. Lower scores indicate improvement.

SECONDARY OUTCOMES:
Stool microbiota changes as assessed by the Dysbiosis index (DI) | 3 months.
  DI is a 5-point scale: DI 1-2: non-dysbiosis, DI: moderate, DI 4-5: severe dysbiosis). Higer scores indicate improvement.

OTHER OUTCOMES:
Adverse events | up to the end point (3 months)
  Patients are encouraged to keep a diary of any adverse events such as diarrhea, constipation, abdominal pain/ if any.

CONTACTS AND LOCATIONS:
Overall Officials: Haldis Lier, MD, PhD, Study Director — Head of Research Department at Helse Finna HF
Locations (1):
- Helse Fonna, Haugesund, Norway

IPD SHARING:
Plan to Share IPD: No
All data are stored at Helse Vest server. Anonymous patients data is available to other research on demand.

REFERENCES:
- [Derived] El-Salhy M, Valeur J, Bronstad I, Gilja OH, Hatlebakk JG. Possible Role of Butyric Acid in Long-Term Symptom Relief in Irritable Bowel Syndrome Patients Following Fecal Microbiota Transplantation. Neurogastroenterol Motil. 2025 Dec;37(12):e70115. doi: 10.1111/nmo.70115. Epub 2025 Aug 1. PMID 40751371
- [Derived] El-Salhy M, Winkel R, Casen C, Hausken T, Gilja OH, Hatlebakk JG. Efficacy of Fecal Microbiota Transplantation for Patients With Irritable Bowel Syndrome at 3 Years After Transplantation. Gastroenterology. 2022 Oct;163(4):982-994.e14. doi: 10.1053/j.gastro.2022.06.020. Epub 2022 Jun 14. PMID 35709830
- [Derived] El-Salhy M, Mazzawi T, Hausken T, Hatlebakk JG. The fecal microbiota transplantation response differs between patients with severe and moderate irritable bowel symptoms. Scand J Gastroenterol. 2022 Sep;57(9):1036-1045. doi: 10.1080/00365521.2022.2064725. Epub 2022 Apr 29. PMID 35486073
- [Derived] El-Salhy M, Mazzawi T, Hausken T, Hatlebakk JG. Irritable bowel syndrome patients who are not likely to respond to fecal microbiota transplantation. Neurogastroenterol Motil. 2022 Sep;34(9):e14353. doi: 10.1111/nmo.14353. Epub 2022 Mar 18. PMID 35302268
- [Derived] El-Salhy M, Kristoffersen AB, Valeur J, Casen C, Hatlebakk JG, Gilja OH, Hausken T. Long-term effects of fecal microbiota transplantation (FMT) in patients with irritable bowel syndrome. Neurogastroenterol Motil. 2022 Jan;34(1):e14200. doi: 10.1111/nmo.14200. Epub 2021 Jun 18. PMID 34145677
- [Derived] El-Salhy M, Valeur J, Hausken T, Gunnar Hatlebakk J. Changes in fecal short-chain fatty acids following fecal microbiota transplantation in patients with irritable bowel syndrome. Neurogastroenterol Motil. 2021 Feb;33(2):e13983. doi: 10.1111/nmo.13983. Epub 2020 Sep 17. PMID 32945066
- [Derived] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769